CLINICAL TRIAL: NCT03089593
Title: Double-blind Placebo-controlled Clinical Trial of Thermogenic Effect of Ginger (Zingiber Officinale) in Eutrophic Women
Brief Title: Thermogenic Effect of Ginger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Adaliene Versiani M. Ferreira, Principal Investigator, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: UFMG 30409114.8.0000.5149
Record Dates: First submitted 2017-03-08; First posted 2017-03-24 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Healthy Volunteers
Keywords: Thermic Effect of Food; Energy Expenditure; Ginger
MeSH Terms: interventions — Cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extract of ginger (Experimental): Healthy and eutrophic women will receive two capsules of 200 mg of ginger extract (5% gingerols) to be taken along with a standardized breakfast.
  Interventions: Other: Extract of ginger
- Cellulose (Placebo Comparator): Healthy and eutrophic women will receive two capsules of 200 mg of placebo (cellulose) to be taken along with a standardized breakfast.
  Interventions: Other: Placebo (Cellulose)

INTERVENTIONS:
Other: Extract of ginger — The volunteers will receive two capsules containing 200mg of extract of ginger with 5% of gingerols (20 mg). Breakfast will be offered (bread, butter, turkey ham and industrialized fruit juice) and the participants will have 15 minutes to eat it.
  Arms: Extract of ginger
Other: Placebo (Cellulose) — The volunteers will receive two capsules containing cellulose (placebo). Breakfast will be offered (bread, butter, turkey ham and industrialized fruit juice) and the participants will have 15 minutes to eat it.
  Arms: Cellulose

SUMMARY:
The main objective of the study is to evaluate the thermogenic effect of ginger.

DETAILED DESCRIPTION:
Healthy and eutrophic women will receive capsules of 200 mg of ginger extract (5% active ingredient) or placebo (cellulose), along with a standardized breakfast, with a minimum seven days washout period.

ELIGIBILITY:
Inclusion Criteria:

* Females;
* Aged between 18 and 60 years old;
* Body mass index between 18.5 and 24.9 kg/m²;
* Agree to sign the informed consent.

Exclusion Criteria:

* Any chronic health conditions (e.g. diabetes, hypertension, chronic renal failure, heart and liver disease);
* Previous operation for weight loss;
* Medications known to affect total energy expenditure;
* Pregnancy and breast-feeding;
* Smoking;
* Alcohol use (>2 doses/day).

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Change in postprandial energy expenditure | Baseline and thereafter at 30, 60, 120, 180 and 240 minutes postprandial
  Energy expenditure will be assessed by indirect calorimetry

SECONDARY OUTCOMES:
Change in oxygen consumption | Baseline and thereafter at 30, 60, 120, 180 and 240 minutes postprandial
  Oxygen consumption will be assessed by indirect calorimetry
Change in blood pressure | Baseline and thereafter at 30, 60, 120, 180 and 240 minutes postprandial
  Blood pressure will be assessed using digital sphygmomanometer
Change in axillary temperature | Baseline and thereafter at 30, 60, 120, 180 and 240 minutes postprandial
  Axillary temperature will be assessed using a digital thermometer
Change in metabolic profile | Baseline and thereafter at 30, 60, 120 and 240 minutes postprandial
  Total cholesterol
Change in heart rate | Baseline and thereafter at 30, 60, 120, 180 and 240 minutes postprandial
  Heart rate will be assessed using digital sphygmomanometer
Change in metabolic profile | Baseline and thereafter at 30, 60, 120 and 240 minutes postprandial
  Glucose levels
Change in metabolic profile | Baseline and thereafter at 30, 60, 120 and 240 minutes postprandial
  HDL-cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela BP Fagundes, Study Chair — Federal University of Minas Gerais
Locations (1):
- Hospital das Clínicas, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fagundes GBP, Rodrigues AMDS, Martins LB, Monteze NM, Correia MITD, Teixeira AL, Ferreira AVM. Acute effects of dry extract of ginger on energy expenditure in eutrophic women: A randomized clinical trial. Clin Nutr ESPEN. 2021 Feb;41:168-174. doi: 10.1016/j.clnesp.2020.10.001. Epub 2020 Nov 9. PMID 33487261